CLINICAL TRIAL: NCT06476821
Title: A Phase 1 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Doses of BMS-986435 (MYK-224) in Healthy Chinese Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, Drug Levels, and Drug Effects of Single Doses of BMS-986435 (MYK-224) in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV029-1010
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: BMS-986435
- Arm 2 (Experimental)
  Interventions: Drug: BMS-986435

INTERVENTIONS:
Drug: BMS-986435 — Specified dose on specified days
  Other Names: MYK-224

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics following a single oral dose of BMS-986435 in healthy adult Chinese participants.

ELIGIBILITY:
Inclusion Criteria:

* Body weight of ≥ 50 kg and body mass index between 18.0 and 28.0 kg/m2, inclusive, at screening.
* Participants must be Chinese (both biological parents are ethnically Chinese).
* Participant has documented LVEF ≥ 60% (2D biplane Simpson's Method) at screening as determined by the echocardiographic core laboratory.

Exclusion Criteria:

* Any acute or chronic medical illness.
* Head injury in the last 2 years, intracranial tumor, or aneurysm.
* History of malignancy of any type, except in situ cervical cancer > 5 years prior to the screening visit or surgically excised nonmelanomatous skin cancers > 2 years prior to the screening visit.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-06-27 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration (Cmax) | Up to Day 30
Time of maximum observed concentration (Tmax) | Up to Day 30
Area under the concentration time curve from time zero to the time of the last quantifiable concentration (AUC(0-T)) | Up to Day 30

SECONDARY OUTCOMES:
Number of participants with Adverse Events | From date of written consent up to 28 days post last dose
Number of participants with Serious Adverse Events | From date of written consent up to 28 days post last dose
Number of participants with AEs leading to discontinuation | From date of written consent up to 28 days post last dose
Number of participants with vital sign abnormalities | Up to Day 31
Number of participants with electrocardiogram (ECG) abnormalities | Up to Day 31
Number of participants with echocardiogram abnormalities | Up to Day 30
Number of participants with physical examination abnormalities | Up to Day 31
Number of participants with clinical laboratory abnormalities | Up to Day 31
Echocardiographic measures of cardiac systolic function: left ventricular ejection fraction (LVEF) | Up to Day 30
Echocardiographic measures of cardiac systolic function: left ventricular outflow tract velocity time integral (LVOT-VTI) | Up to Day 30
Echocardiographic measures of cardiac systolic function: left ventricular fractional shortening (LVFS) | Up to Day 30
Echocardiographic measures of cardiac systolic function: left ventricular global longitudinal strain (LV GLS) | Up to Day 30
Echocardiographic measures of cardiac systolic function: left ventricle stroke volume (LVSV) | Up to Day 30
Echocardiographic measures of cardiac diastolic function: lateral early diastolic mitral annular velocity (e') | Up to Day 30
Echocardiographic measures of cardiac diastolic function: septal e' | Up to Day 30
Echocardiographic measures of cardiac diastolic function: early diastolic mitral inflow velocity to early diastolic mitral annular velocity (E/e') | Up to Day 30
Echocardiographic measures of cardiac diastolic function: early diastolic mitral inflow velocity to late diastolic mitral inflow velocity ratio (E/A ratio) | Up to Day 30
Echocardiographic measures of cardiac structure: LV mass index | Up to Day 30
Echocardiographic measures of cardiac structure: LV atrial volume index | Up to Day 30
Echocardiographic measures of cardiac structure: interventricular septal thickness | Up to Day 30
Echocardiographic measures of cardiac structure: posterior wall thickness | Up to Day 30
Echocardiographic measures of cardiac structure: LV end diastolic volume | Up to Day 30
Echocardiographic measures of cardiac structure: LV end systolic volume | Up to Day 30
Echocardiographic measures of cardiac structure: LV end systolic volume index | Up to Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Xuhui District, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com